CLINICAL TRIAL: NCT00872989
Title: Randomized Phase II Study of Docetaxel Followed by Vandetanib (ZD6474) vs. Docetaxel Plus Vandetanib in Patients With Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: S0904: Docetaxel With or Without Vandetanib in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000638595; S0904 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent fallopian tube cancer; recurrent primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who progress also receive oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of a second disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: vandetanib
- Arm II (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: vandetanib

INTERVENTIONS:
Drug: docetaxel — Given IV
Drug: vandetanib — Given orally

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether docetaxel is more effective when given alone or together with vandetanib.

PURPOSE: This randomized phase II trial is studying docetaxel given together with or without vandetanib to see how well it works in treating patients with persistent or recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the clinical efficacy of docetaxel and vandetanib relative to docetaxel alone in patients with platinum-resistant, recurrent, refractory, or progressive/persistent ovarian epithelial, primary peritoneal, or fallopian tube cancer, as measured by progression-free survival.
* To evaluate the response rate (complete and partial) and duration of overall survival of these patients.
* To evaluate the response (complete and partial) and time to treatment failure after treatment with single agent vandetanib following progression on single agent docetaxel.
* To evaluate the frequency and severity of adverse events as assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0.
* To evaluate the toxicity of single agent vandetanib following docetaxel as assessed by CTCAE v4.0.

OUTLINE: Patients are stratified according to prior treatment with antiangiogenesis agents (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who progress also receive oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of a second disease progression or unacceptable toxicity.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1 and oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal carcinoma

  * Recurrent, refractory, or progressive/persistent disease
* Measurable or non-measurable disease documented by CT scan of the abdomen and pelvis
* Must have received 1 prior platinum-based chemotherapy regimen for management of primary disease containing carboplatin, cisplatin, or other organoplatinum compound

  * Initial treatment may have included any of the following:

    * High-dose therapy
    * Consolidation therapy
    * Non-cytotoxic agent therapy
    * Extended therapy administered after surgical or non-surgical assessment
  * Additional cytotoxic regimen for recurrent, refractory, or progressive/persistent disease, including re-treatment with primary treatment regimen
* No more than 3 prior regimens for recurrent, refractory, persistent, or progressive disease.

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mcl
* Platelet count ≥ 100,000/mcl
* Serum creatinine normal OR calculated creatinine clearance ≥ 30 mL/min
* Urine protein:creatinine ratio < 1
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* aspartate aminotransferase - alanine aminotransferase (AST or ALT) ≤ 2.5 times ULN (≤ 5 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of vandetanib therapy
* No neuropathy ≥ grade 2 CTCAE v4.0
* No active infection requiring systemic or intravenous antibiotics
* No significant traumatic injury within the past 28 days
* No significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension (i.e., systolic blood pressure [BP] > 140 mm Hg or diastolic BP > 90 mm Hg) within the past 28 days
  * Myocardial infarction superior vena cava syndrome, or New York Heart Association (NYHA) class II-IV heart disease within the past 3 months
  * Presence of left bundle branch block
  * Congenital long QT syndrome or first degree relative with unexplained sudden death < 40 years of age
  * QT interval with Bazett's correction that is unmeasurable or ≥ 480 msec by screening ECG
  * History of symptomatic arrhythmia (i.e., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) requiring treatment (≥ CTCAE grade 3) or asymptomatic sustained ventricular tachycardia

    * Atrial fibrillation controlled on medication allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy (except alopecia) to NCI CTCAE v3.0 grade ≤ 1
* No prior vandetanib

  * Treatment with other anti-vascular endothelial growth factor (VEGF) targeted therapy allowed
* No prior docetaxel or any non-cytotoxic therapy (excluding hormonal therapy) for recurrent disease, regardless of whether it was part of primary treatment

  * Prior docetaxel as part of front-line cytotoxic regimen (including maintenance therapy) allowed as long as no disease progression on or within 6 months after receiving docetaxel
* At least 7 days since prior hormonal therapy for the malignant tumor

  * Concurrent hormone replacement therapy for menopausal symptoms allowed
* At least 28 days since other prior therapy for the malignant tumor, including immunologic agents
* More than 7 days since prior minor surgical procedures, fine needle aspirates, or core biopsies
* More than 14 days since prior and no concurrent potent inducers of cytochrome P450 3A4 (CYP3A4) function
* More than 14 days since prior and no concurrent medications having a risk of causing Torsades de Pointes or risk of QTc prolongation

  * Patients receiving a drug that has a risk of QTc prolongation must not have QTc ≥ 460 msec
* More than 28 days since prior investigational agents for any purpose
* More than 28 days since prior and no concurrent major surgical procedure or open biopsy
* More than 5 years since prior chemotherapy for abdominal or pelvic tumor, except treatment of ovarian, fallopian tube, or primary peritoneal cancer

  * Prior adjuvant chemotherapy for localized breast cancer allowed, provided it was completed more than 3 years prior to study, and the patient remains free of recurrent or metastatic disease
* More than 5 years since prior radiotherapy to any portion of the abdominal cavity or pelvis, except for the treatment of ovarian, fallopian tube, or primary peritoneal cancer

  * Prior radiotherapy for localized cancer of the breast, head and neck, or skin allowed, provided it was completed more than 3 years prior to study, and the patient remains free of recurrent or metastatic disease
  * No prior radiation to more than 25% of marrow-bearing areas

    * More than 28 days since prior radiotherapy
* No other concurrent investigational or commercial agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-03; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Coleman, MD, Study Chair — M.D. Anderson Cancer Center
Locations (137):
- United States (137):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - NEA Medical Center - Stadium Boulevard, Jonesboro, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center, Vallejo, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Coleman RL, Moon J, Sood AK, Hu W, Delmore JE, Bonebrake AJ, Anderson GL, Chambers SK, Markman M. Randomised phase II study of docetaxel plus vandetanib versus docetaxel followed by vandetanib in patients with persistent or recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma: SWOG S0904. Eur J Cancer. 2014 Jun;50(9):1638-48. doi: 10.1016/j.ejca.2014.03.005. Epub 2014 Apr 4. PMID 24709487
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Docetaxel: Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who progress also receive oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of a second disease progression or unacceptable toxicity.
  docetaxel: Given IV
  vandetanib: Given orally
- Arm II: Docetaxel + Vandetanib: Patients receive docetaxel IV over 1 hour on day 1 and oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  docetaxel: Given IV
  vandetanib: Given orally
Period: Overall Study
Arm/Group | Arm I: Docetaxel | Arm II: Docetaxel + Vandetanib
Started | 66 | 63
Completed | 1 | 0
Not Completed | 65 | 63
Not completed — Adverse Event | 7 | 15
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Progression/relapse | 47 | 35
Not completed — Not protocol specified | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Docetaxel | Arm II: Docetaxel + Vandetanib | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Continuous [Median (Full Range); unit: years] | 61.7 [32.6 to 80] | 61.9 [34.3 to 82.5] | 61.9 [32.6 to 82.5]
Gender [Count of Participants; unit: Participants]
  Female | 66 | 63 | 129
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 58 | 56 | 114
  Black | 4 | 4 | 8
  Asian | 4 | 2 | 6
  Unknown | 0 | 1 | 1
Hispanic [Number; unit: participants]
  Yes | 2 | 4 | 6
  No | 64 | 58 | 122
  Unknown | 0 | 1 | 1
Prior Antiangiogenic Therapy [Number; unit: participants]
  Yes | 12 | 9 | 21
  No | 54 | 54 | 108
Primary Site [Number; unit: participants]
  Fallopian Tube | 3 | 4 | 7
  Ovary | 56 | 53 | 109
  Peritoneal | 7 | 6 | 13
Performance Status [Number; unit: participants] — Patients performance status (PS) are graded into five grades. In this trial, only patients with PS 0-2 are included. The criteria for each grade are the followings:
  0: Fully active, able to carry on all pre-disease performance without restriction;
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work;
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  participants
    0 | 37 | 33 | 70
    1 | 27 | 26 | 53
    2 | 2 | 4 | 6
Baseline serum level of cancer-antigen 125 (CA-125) [Number; unit: participants] — The cutoff point for CA-125 is 35 units/mL. Anything above 35 units/mL is abnormal.
  participants
    ≤ 35 units/mL | 17 | 10 | 27
    > 35 units/mL | 49 | 53 | 102
Prior treatment with platinum for recurrent disease [Number; unit: participants] | 34 | 28 | 62

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Disease assessments were performed every 6 weeks for as long as the patient remained on protocol, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Docetaxel | Arm II: Docetaxel + Vandetanib
Number analyzed (Participants) | 66 | 63
months | 3.5 [2.3 to 4.6] | 3.0 [1.6 to 4.3]
Statistical Analysis 1: Comparison: Arm I: Docetaxel vs Arm II: Docetaxel + Vandetanib; Test type: Superiority or Other; p = 0.49, Regression, Cox; Hazard Ratio (HR) = 0.99, 80% CI 2-sided [0.79 to 1.26]

2. Secondary Outcome: Number of Participants With a Complete Response, Partial Response, Stable Disease, or Increasing Disease
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR in conjunction with measured CA125 responses
Time Frame: Disease assessment for responses were performed every 6 weeks for as long as the patient remained on protocol treatment, up to 5 years.
Population: Analysis of response is in the subset of patients who had at least one measurable target lesion at baseline.
Measure: Number; unit: participants
Arm/Group | Arm I: Docetaxel | Arm II: Docetaxel + Vandetanib
Number analyzed (Participants) | 57 | 52
participants
  Complete Response | 0 | 0
  Partial Response | 5 | 6
  Unconfirmed Complete Response | 1 | 0
  Unconfirmed Partial Response | 2 | 2
  Stable/No Response | 19 | 17
  Increasing Disease | 23 | 20
  Symptomatic Deterioration | 0 | 1
  Assessment Inadequate | 7 | 6

3. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: every 3 months for two years and then every 6 months for 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Docetaxel | Arm II: Docetaxel + Vandetanib
Number analyzed (Participants) | 66 | 63
months | 18 [13.7 to 26.1] | 14 [9.9 to 19.7]
Statistical Analysis 1: Comparison: Arm I: Docetaxel vs Arm II: Docetaxel + Vandetanib; Test type: Superiority or Other; p = 0.83, Regression, Cox; Hazard Ratio (HR) = 1.25, 80% CI 2-sided [0.93 to 1.68]

4. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 3.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment was evaluated before each treatment cycle (21 days), up to 5 years.
Population: Eligible patients who had received the protocol treatments were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Docetaxel | Docetaxel + Vandetanib | Vandetanib
Number analyzed (Participants) | 64 | 61 | 33
Participants
  Abdominal pain | 0 | 1 | 0
  Allergic reaction | 0 | 1 | 0
  Anemia | 1 | 2 | 0
  Anorexia | 1 | 2 | 1
  Ascites | 0 | 0 | 1
  Bladder infection | 0 | 1 | 0
  Chest pain - cardiac | 0 | 1 | 0
  Constipation | 0 | 1 | 0
  Dehydration | 3 | 3 | 0
  Depression | 0 | 0 | 1
  Diarrhea | 2 | 5 | 1
  Dyspnea | 0 | 2 | 1
  Edema limbs | 1 | 0 | 0
  Fatigue | 6 | 5 | 1
  Febrile neutropenia | 0 | 1 | 0
  Gastrointestinal pain | 0 | 1 | 0
  Generalized muscle weakness | 1 | 1 | 0
  Hypercalcemia | 1 | 0 | 0
  Hyperglycemia | 1 | 1 | 0
  Hypertension | 0 | 0 | 2
  Hypocalcemia | 2 | 1 | 0
  Hypokalemia | 1 | 1 | 1
  Hypomagnesemia | 1 | 2 | 0
  Hyponatremia | 1 | 0 | 0
  Hypotension | 1 | 0 | 0
  Hypoxia | 0 | 1 | 0
  Leukocytosis | 1 | 1 | 0
  Lung infection | 2 | 0 | 0
  Lymphocyte count decreased | 0 | 1 | 0
  Mucositis oral | 1 | 1 | 0
  Myalgia | 0 | 0 | 1
  Nail infection | 0 | 1 | 0
  Nausea | 5 | 2 | 1
  Neutrophil count decreased | 32 | 28 | 0
  Palmar-plantar erythrodysesthesia syndrome | 1 | 0 | 0
  Papulopustular rash | 0 | 1 | 0
  Peripheral sensory neuropathy | 3 | 0 | 0
  Platelet count decreased | 0 | 1 | 0
  Pneumonitis | 0 | 1 | 0
  Pruritus | 0 | 1 | 0
  Rash acneiform | 0 | 1 | 0
  Rash maculo-papular | 0 | 4 | 0
  Sinus bradycardia | 0 | 1 | 0
  Skin and subcutaneous tissue disorders - Other | 0 | 1 | 0
  Stoma site infection | 0 | 1 | 0
  Thromboembolic event | 0 | 1 | 0
  Treatment related secondary malignancy | 0 | 1 | 0
  Urinary tract infection | 0 | 2 | 0
  Vomiting | 3 | 3 | 1
  White blood cell decreased | 20 | 20 | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure after treatment with single agent vandetanib following progression on single agent docetaxel. Disease assessments were performed every 6 weeks for as long as the patient remained on protocol, up to 5 years.
Time Frame: Disease assessments were performed every 6 weeks for as long as the patient remained on protocol, up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Vandetanib: Vandetanib treated patients
Arm/Group | Vandetanib
Number analyzed (Participants) | 33
Months | 1.4 [1.3 to 1.6]

6. Secondary Outcome: Number of Participants With a Complete Response, Partial Response, Stable Disease, or Increasing Disease After Treatment With Single Agent Vandetanib Following Progression on Single Agent Docetaxel
Description: as for outcome 2
Time Frame: Disease assessments were performed every 6 weeks for as long as the patient remained on protocol, up to 5 years.
Population: Analysis of response is in the subset of patients who had at least one measurable target lesion at baseline.
Measure: Number; unit: participants
Groups:
- Vandetanib: Patients elected to participant in the crossover registration in Vandetanib after progression in single agent docetaxel.
Arm/Group | Vandetanib
Number analyzed (Participants) | 30
participants
  Complete Response | 0
  Partial Response | 0
  Unconfirmed Complete Response | 0
  Unconfirmed Partial Response | 1
  Stable/No Response | 8
  Increasing Disease | 20
  Assessment Inadequate | 1

ADVERSE EVENTS:
Time Frame: Toxicity assessments was evaluated before each treatment cycle (21 days), up to 5 years.
Groups:
- Docetaxel; Docetaxel + Vandetanib; Vandetanib: Adverse events are analyzed in the subset of patients who received at least one dose of drug.
Arm/Group | Docetaxel | Docetaxel + Vandetanib | Vandetanib
Serious Adverse Events (participants affected / at risk) | 1/64 | 31/61 | 7/33
Other Adverse Events (participants affected / at risk) | 61/64 | 59/61 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=64) | Docetaxel + Vandetanib (N=61) | Vandetanib (N=33)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 3
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2
Death NOS (General disorders) | 0 | 2 | 1
Fatigue (General disorders) | 0 | 2 | 1
General disorders and admin site conditions - Other (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 19 | 0
White blood cell decreased (Investigations) | 0 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=64) | Docetaxel + Vandetanib (N=61) | Vandetanib (N=33)
Anemia (Blood and lymphatic system disorders) | 47 | 27 | 11
Palpitations (Cardiac disorders) | 0 | 4 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 2
Watering eyes (Eye disorders) | 5 | 7 | 1
Abdominal distension (Gastrointestinal disorders) | 10 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 16 | 19 | 10
Ascites (Gastrointestinal disorders) | 4 | 4 | 1
Bloating (Gastrointestinal disorders) | 1 | 4 | 1
Constipation (Gastrointestinal disorders) | 25 | 23 | 12
Diarrhea (Gastrointestinal disorders) | 27 | 26 | 13
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 2
Mucositis oral (Gastrointestinal disorders) | 21 | 19 | 1
Nausea (Gastrointestinal disorders) | 34 | 30 | 8
Vomiting (Gastrointestinal disorders) | 19 | 14 | 4
Chills (General disorders) | 2 | 5 | 0
Edema limbs (General disorders) | 14 | 10 | 3
Fatigue (General disorders) | 47 | 39 | 18
Fever (General disorders) | 5 | 5 | 0
Pain (General disorders) | 4 | 5 | 2
Alanine aminotransferase increased (Investigations) | 4 | 8 | 2
Alkaline phosphatase increased (Investigations) | 7 | 12 | 7
Aspartate aminotransferase increased (Investigations) | 4 | 7 | 4
Creatinine increased (Investigations) | 5 | 12 | 8
Lymphocyte count decreased (Investigations) | 1 | 5 | 1
Neutrophil count decreased (Investigations) | 35 | 25 | 1
Platelet count decreased (Investigations) | 7 | 8 | 0
Weight loss (Investigations) | 3 | 1 | 3
White blood cell decreased (Investigations) | 34 | 25 | 2
Anorexia (Metabolism and nutrition disorders) | 18 | 16 | 8
Dehydration (Metabolism and nutrition disorders) | 6 | 6 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 13 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 10 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 11 | 1
Hypokalemia (Metabolism and nutrition disorders) | 11 | 6 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 25 | 7
Hyponatremia (Metabolism and nutrition disorders) | 7 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 16 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 3 | 2
Dizziness (Nervous system disorders) | 8 | 5 | 1
Dysgeusia (Nervous system disorders) | 7 | 5 | 0
Headache (Nervous system disorders) | 6 | 8 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 34 | 24 | 13
Anxiety (Psychiatric disorders) | 5 | 7 | 1
Depression (Psychiatric disorders) | 6 | 4 | 2
Insomnia (Psychiatric disorders) | 13 | 9 | 4
Hematuria (Renal and urinary disorders) | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 12 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 43 | 36 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 6 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 9 | 8 | 1
Nail loss (Skin and subcutaneous tissue disorders) | 5 | 3 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 6 | 3 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 9 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 14 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 23 | 0
Hot flashes (Vascular disorders) | 5 | 0 | 1
Hypertension (Vascular disorders) | 1 | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less